CLINICAL TRIAL: NCT02038764
Title: A Phase 1 Study To Evaluate The Safety, Tolerability, Immunogenicity, Pharmacokinetics And Pharmacodynamics Of Multiple Ascending Doses Of Pf-06342674 (rn168) In Adults With Type 1 Diabetes
Brief Title: A Study To Assess The Safety Of PF-06342674 In Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Basic Science
Other Study IDs: B4351003
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Phase 1; RN168; Adults; Type 1 Diabetes; T1D
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- PF-06342674 (Experimental)
  Interventions: Biological: PF-06342674 Dose A; Biological: PF-06342674 Dose B; Biological: PF-06342674 Dose C; Biological: PF-06342674 Dose D

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Biological: PF-06342674 Dose A — Multiple SC Doses
  Arms: PF-06342674
Biological: PF-06342674 Dose B — Multiple SC Doses
  Arms: PF-06342674
Biological: PF-06342674 Dose C — Multiple SC Doses
  Arms: PF-06342674
Biological: PF-06342674 Dose D — Multiple SC Doses
  Arms: PF-06342674

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of multiple doses of PF-06342674. Several dose levels will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women and men age 18 and older.
* Diagnosis of type 1 diabetes within 2 years of randomization.
* Peak stimulated C-peptide levels ≥ 0.15 ng/mL.

Exclusion Criteria:

* Anticipated ongoing use of diabetes medications other than insulin.
* Evidence or history of diabetic complications with significant end-organ damage.
* Episode of severe hypoglycemia within 60 days of randomization.
* Multiple hospitalizations for diabetic ketoacidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (21):
  - VA San Diego Healthcare System (Drug Shipment), San Diego, California
  - Veterans Administration San Diego Healthcare System, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Barbara Davis Center, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Yale New Haven Hospital - Investigational Drug Services, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Duchossois Center for Advanced Medicine, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago Clinical Resource Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University Of Minnesota Fairview Pharmacy Services, Minneapolis, Minnesota
  - University Of Minnesota Medical School, Minneapolis, Minnesota
  - Barnes- Jewish HOSP Att: Kathryn Vehe, St Louis, Missouri
  - Washington University - Center for Advanced Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Duke Clinical Research Unit, Durham, North Carolina
  - Duke University Health Systems (DUHS) Investigational Drug Services, Durham, North Carolina

REFERENCES:
- [Derived] Herold KC, Bucktrout SL, Wang X, Bode BW, Gitelman SE, Gottlieb PA, Hughes J, Joh T, McGill JB, Pettus JH, Potluri S, Schatz D, Shannon M, Udata C, Wong G, Levisetti M, Ganguly BJ, Garzone PD; RN168 Working Group. Immunomodulatory activity of humanized anti-IL-7R monoclonal antibody RN168 in subjects with type 1 diabetes. JCI Insight. 2019 Dec 19;4(24):e126054. doi: 10.1172/jci.insight.126054. PMID 31852846
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4351003&StudyName=A%20Study%20To%20Assess%20The%20Safety%20Of%20PF-06342674%20In%20Adults%20With%20Type%201%20Diabetes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 37 participants were assigned to study treatment (placebo: 7 subjects; PF-06342674: 30 subjects)
Groups:
- Placebo: Participants were randomly assigned to placebo in a 2/8 ratio in Cohorts 1 through 3 and a 1/4 ratio in Cohort 4. The treatment was given as a subcutaneous injection(s)
- PF-06342674 1 mg/kg; PF-06342674 3 mg/kg; PF-06342674 8 mg/kg: Participants received their dose as a subcutaneous injection(s) once every two weeks (q2w) up to 6 doses.
- PF-06342674 6 mg/kg: Participants received their dose as a subcutaneous injection(s) once a week (q1w) up to 12 doses.
Period: Overall Study
Arm/Group | Placebo | PF-06342674 1 mg/kg | PF-06342674 3 mg/kg | PF-06342674 6 mg/kg | PF-06342674 8 mg/kg
Started | 7 | 8 | 9 | 5 | 8
Completed | 6 | 7 | 7 | 5 | 7
Not Completed | 1 | 1 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Other | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06342674 1 mg/kg | PF-06342674 3 mg/kg | PF-06342674 6 mg/kg | PF-06342674 8 mg/kg | Total
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (11.1) | 25.6 (8.5) | 37.8 (15.8) | 29 (12.3) | 30.8 (7.7) | 31.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 6 | 0 | 4 | 15
  Male | 5 | 5 | 3 | 5 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting or Intolerable Treatment Related Adverse Events (AEs)
Description: Number of participants with dose limiting or intolerable treatment related adverse events (AEs) was reported. An AE was any untoward medical occurrence in a clinical investigation subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage.
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Cohort 1 PF-06342674 1 mg/kg; Cohort 2 PF-06342674 3 mg/kg; Cohort 3 PF-06342674 8 mg/kg: Participants received their dose as a subcutaneous injection(s) once every two weeks (q2w) up to 6 doses.
- Cohort 4 PF-06342674 6 mg/kg: Participants received their dose as a subcutaneous injection(s) once a week (q1w) up to 12 doses.
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With All-Causality Treatment Emergent Adverse Events(TEAEs)
Description: Number of participants with all-causality treatment emergent adverse events were reported. An AE was any untoward medical occurrence in a clinical investigation subject administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. TEAEs were those AEs with initial onset or increasing in severity after the first dose of study drug. TEAEs included both serious and non-serious AE
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants | 7 | 8 | 7 | 5 | 6

3. Primary Outcome: Number of Participants With Treatment-Related TEAEs
Description: Number of participants with treatment-related TEAEs were reported. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An AE was any untoward medical occurrence in a clinical investigation subject administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. TEAEs were those AEs with initial onset or increasing in severity after the first dose of study drug.
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants | 5 | 6 | 6 | 4 | 5

4. Primary Outcome: Number of Participants With All-Causality TEAEs Listed by Common Terminology Criteria for Adverse Events (CTCAE) Grade
Description: TEAEs were those AEs with initial onset or increasing in severity after the first dose of study drug. CTCAE version 4.03 was used to grade the severity of TEAEs. Grade 1 referred to mild AEs; Grade 2 referred to moderate AEs; Grade 3 referred to severe AEs; Grade 4 referred to AEs with life-threatening consequences, and urgent intervention was needed to manage them; Grade 5 referred to death related to AE.
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants
  Grade 1 | 3 | 2 | 1 | 3 | 1
  Grade 2 | 2 | 6 | 4 | 0 | 4
  Grade 3 | 2 | 0 | 2 | 2 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With All-Causality Treatment-Emergent Hypoglycemic Adverse Events
Description: Number of participants with all-causality treatment-emergent hypoglycemic adverse events was reported. Any blood glucose values less than(<)55 mg/dL with or without symptoms was reported as adverse events of hypoglycemia.
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants | 4 | 4 | 5 | 1 | 3

6. Primary Outcome: Number of Participants With All-Causality Treatment-Emergent Hypoglycemic Adverse Events Listed by CTCAE Grade
Description: Any blood glucose values <55 mg/dL with or without symptoms was reported as adverse events of hypoglycemia. CTCAE version 4.03 was used to grade the severity of TEAEs. Grade 1 referred to mild AEs; Grade 2 referred to moderate AEs; Grade 3 referred to severe AEs; Grade 4 referred to AEs with life-threatening consequences, and urgent intervention was needed to manage them; Grade 5 referred to death related to AE.
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants
  Grade 1 | 1 | 0 | 1 | 0 | 0
  Grade 2 | 1 | 4 | 3 | 0 | 2
  Grade 3 | 2 | 0 | 1 | 1 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: The following laboratory test parameters were evaluated in this study: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, absolute total neutrophils, absolute eosinophils, absolute basophils, absolute monocytes, and absolute lymphocytes),coagulation (partial thromboplastin time, prothrombin, and prothrombin international ratio), liver function(total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, total protein, and albumin), renal function (blood urea nitrogen, creatinine, and uric acid), electrolytes (sodium, potassium, chloride, calcium, and venous bicarbonate), clinical chemistry(glucose, glycosylated, and hemoglobin), and urinalysis (pH, qualitative glucose, qualitative protein, qualitative blood, urobilinogen, qualitative bilirubin, nitrites, leukocyte, esterase and microscopy).
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants | 7 | 7 | 8 | 5 | 7

8. Primary Outcome: Number of Participants With Vital Signs That Met the Criteria for Potential Clinical Concern(Absolute Values)
Description: Number of participants with vital signs data of absolute values meeting criteria of potential clinical concern. Absolute values were analyzed for systolic blood pressure (SBP), diastolic blood pressure (DBP), and pulse rate. Number of participants with vital signs data meeting the following criteria was reported: Criterion A: SBP <90 millimeter of mercury(mmHg); Criterion B: DBP <50 mmHg; Criterion C: pulse rate < 40 beats per minute(BPM); Criterion D: pulse rate >120 BPM
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants
  Criterion A | 0 | 0 | 1 | 0 | 0
  Criterion B | 1 | 0 | 0 | 0 | 0
  Criterion C | 1 | 0 | 0 | 0 | 0
  Criterion D | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Vital Signs That Met the Criteria for Potential Clinical Concern(Decreases From Baseline)
Description: The number of participants with vital signs data of maximum decrease from baseline meeting the following criteria was reported: Criterion A: maximum decrease from baseline in systolic BP >= 30 mmHg; Criterion B: maximum decrease from baseline in diastolic BP >=20 mmHg
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants
  Criterion A | 0 | 0 | 0 | 0 | 0
  Criterion B | 0 | 0 | 0 | 0 | 1

10. Primary Outcome: Number of Participants With Vital Signs That Met the Criteria for Potential Clinical Concern(Increases From Baseline)
Description: The number of participants with vital signs data of maximum increase from baseline meeting the following criteria was reported: Criterion A: maximum increase from baseline in systolic BP >= 30 mmHg; Criterion B: maximum increase from baseline in diastolic BP >= 20 mmHg
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants
  Criterion A | 0 | 0 | 0 | 1 | 0
  Criterion B | 1 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Electrocardiogram(ECG) Data That Met the Criteria for Potential Clinical Concern(Absolute Value)
Description: The number of participants with ECG absolute values meeting the following criteria was reported: Criterion A: maximum PR interval (time from the beginning of P wave to the start of QRS complex, corresponding to the end of atrial depolarization and onset of ventricular depolarization) >=300 msec; Criterion B: maximum QRS complex(time from Q wave to the end of S wave, corresponding to ventricle depolarization) >=200 msec; Criterion C: maximum QTcF interval (time from the beginning of Q wave to the end of T wave corresponding to electrical systole, corrected for heart rate using Fridericia's formula) 450-<480 msec; Criterion D: maximum QTcF interval 480-<500 msec; Criterion E: maximum QTcF interval (Fridericia's correction) >=500 msec
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants
  Criterion A | 0 | 0 | 0 | 0 | 0
  Criterion B | 0 | 0 | 0 | 0 | 0
  Criterion C | 1 | 0 | 3 | 1 | 0
  Criterion D | 0 | 0 | 0 | 0 | 0
  Criterion E | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Electrocardiogram(ECG) Data That Met the Criteria for Potential Clinical Concern(Increases From Baseline)
Description: Number of participants with ECG meeting the following criteria was reported: Criterion A: maximum PR interval increase from baseline percentage change (PctChg)>= 25/50%; Criterion B: maximum QRS complex increase from baseline PctChg >= 25/50%; Criterion C: maximum QTcF interval increase from baseline 30<=change<60 msec; Criterion D: maximum QTcF interval increase from baseline change >=60 msec.
Time Frame: Day 1 through Day 127
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants
  Criterion A | 0 | 0 | 0 | 0 | 0
  Criterion B | 0 | 0 | 0 | 0 | 0
  Criterion C | 1 | 0 | 2 | 0 | 1
  Criterion D | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Serum Anti-PF-06342674 Antibody Response Listed by Visit
Description: Number of participants with serum anti-PF-06342674 antibody response to the intramuscular tetanus vaccine was reported. Positive Anti-PF-06342674 Antibody response is defined as anti-tetanus toxoid immunoglobulin G (IgG) titer value >=100
Time Frame: Day 1, Day 15, Day 29, Day 57, Day 85, and Day127 and follow-up visits
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 7 | 8 | 9 | 5 | 8
participants
  Day 1 Negative | 2 | 8 | 9 | 5 | 8
  Day 1 Positive | 0 | 0 | 0 | 0 | 0
  Day 15 Negative | 2 | 6 | 6 | 5 | 8
  Day 15 Positive | 0 | 2 | 2 | 0 | 0
  Day 29 Negative | 2 | 4 | 6 | 5 | 8
  Day 29 Positive | 0 | 4 | 2 | 0 | 0
  Day 57 Negative | 1 | 4 | 4 | 3 | 7
  Day 57 Positive | 0 | 4 | 4 | 2 | 1
  Day 85 Negative | 1 | 3 | 4 | 1 | 4
  Day 85 Positive | 0 | 5 | 3 | 4 | 4
  Day 127 Negative | 1 | 2 | 5 | 0 | 2
  Day 127 Positive | 0 | 6 | 2 | 5 | 6
  Follow-up1 Negative | 0 | 1 | 0 | 0 | 2
  Follow-up1 Positive | 0 | 4 | 3 | 5 | 5
  Follow-up2 Negative | 0 | 3 | 1 | 0 | 3
  Follow-up2 Positive | 0 | 1 | 1 | 5 | 1
  Follow-up3 Negative | 0 | 1 | 0 | 4 | 0
  Follow-up3 Positive | 0 | 1 | 1 | 1 | 1

14. Secondary Outcome: Area Under Concentration-Time Curve From Time Zero to Time Tau(AUCtau) on Day 1 and Day 71
Description: Area under the concentration-time profile from time 0 to time tau (τ), the dosing interval, where tau = 168 hours for once a week dosing; tau = 336 hours for once every 2 weeks dosing. On Day 1, 3 participants in cohort 1 had reportable AUCtau values. On Day 71, 6 participants in cohort 1 and 2 participants in cohort 4 had reportable AUCtau values
Time Frame: 0,1,4 hours post-dose on Day 1 and Day 71
Population: All participants randomized and treated who had at least 1 of the PK parameters of interest were analyzed. On Day 1, 3 participants in cohort 1 had reportable AUCtau values. On Day 71, 6 participants in cohort 1 and 2 participants in cohort 4 had reportable AUCtau values
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 8 | 8 | 5 | 8
ng*hr/mL
  Day 1 | 384900 (43) | 1323000 (43) | 2570000 (31) | 5805000 (28)
  Day 71 | 426700 (58) | 2029000 (29) | NA (NA) — Parameters not reported because less than 3 participants had reportable values, which failed to meet the Pfizer standard that at least 3 subjects must have an adequate dataset available for calculating and reporting PK parameter. | 7869000 (42)

15. Secondary Outcome: Apparent Oral Clearance (CL/F) on Day 71
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. On Day 71, 6 participants in cohort 1 had reportable CL/F values
Time Frame: 0,1,4 hours post-dose on Day 71
Population: All participants randomized and treated who had at least 1 of the PK parameters of interest were analyzed. Day 71, 6 participants in cohort 1 had reportable CL/F values
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 8 | 8 | 2 | 8
mL/hr/kg | 2.340 (58) | 1.477 (29) | NA (NA) — Parameters not reported because less than 3 participants had reportable values, which failed to meet the Pfizer standard that at least 3 subjects must have an adequate dataset available for calculating and reporting PK parameter | 1.017 (42)

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 1 and Day 71
Description: Maximum serum concentration was observed directly from data on Day 1 and Day 71. On Day 71, 2 participants in cohort 4 had reportable Cmax values
Time Frame: 0, 1, 4 hours post-dose on Day 1 and Day 71
Population: All enrolled participants treated who had at least 1 concentration value. On Day 71, 2 participants in cohort 4 had reportable Cmax values
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 8 | 8 | 5 | 8
ng/mL
  Day 1 | 2114 (83) | 8512 (42) | 20890 (29) | 31610 (27)
  Day 71 | 2612 (89) | 10600 (22) | NA (NA) — Parameters not reported because less than 3 participants had reportable values, which failed to meet the Pfizer standard that at least 3 subjects must have an adequate dataset available for calculating and reporting PK parameter | 39870 (34)

17. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 1 and Day 71
Description: Time to reach maximum observed plasma concentration was observed directly from data as time of first occurrence on Day 1 and Day 71. On Day 71, 2 participants in cohort 4 had reportable Tmax values
Time Frame: 0, 1, 4 hours post-dose on Day 1 and Day 71
Population: All participants randomized and treated who had at least 1 of the PK parameters of interest were analyzed.On Day 71, 2 participants in cohort 4 had reportable Tmax values
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 8 | 8 | 5 | 8
hr
  Day 1 | 48.8 (83) [45.9 to 169] | 48.9 (42) [47.4 to 96.8] | 48.1 (29) [46.2 to 73.0] | 51.8 (27) [45.5 to 71.8]
  Day 71 | 48.9 (89) [22.5 to 72.1] | 60.2 (22) [45.8 to 143] | NA (NA) [NA to NA] — Parameters not reported because less than 3 participants had reportable values, which failed to meet the Pfizer standard that at least 3 subjects must have an adequate dataset available for calculating and reporting PK parameter | 86.3 (34) [47.5 to 146]

18. Secondary Outcome: Plasma Decay Half-Life (t1/2) on Day 71
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. On Day 71, 2 participants in cohort 1, 5 participants in cohort 2, and 7 participants in cohort 3 had reportable values for t1/2
Time Frame: 0, 1, 4 hours post-dose on Day 71
Population: All participants randomized and treated who had at least 1 of the PK parameters of interest were analyzed. On Day 71, 2 participants in cohort 1 , 5 participants in cohort 2, and 7 participants in cohort 3 had reportable values for t1/2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 8 | 8 | 2 | 8
hr | NA (NA) — Parameters not calculated because the first post dose was 168 hours (τ). | 64.62 (7.34) | NA (NA) — Parameters not calculated because the first post dose was 168 hours (τ) | 85.54 (23.54)

19. Secondary Outcome: Apparent Volume of Distribution (Vz/F) on Day 71
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed. On Day 71, 1 participant in cohort 1, 5 participants in cohort 2, and 7 participants in cohort 3 had reportable Vz/F values
Time Frame: 0, 1, 4 hours post-dose on Day 71
Population: All participants randomized and treated who had at least 1 of the PK parameters of interest were analyzed. On Day 71, 1 participant in cohort 1, 5 participants in cohort 2, and 7 participants in cohort 3 had reportable Vz/F values
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 8 | 8 | 2 | 8
mL/kg | NA (NA) — Parameters not calculated because the first post dose was 168 hours (τ). | 141.2 (18) | NA (NA) — Parameters not reported because less than 3 participants had reportable values, which failed to meet the Pfizer standard that at least 3 subjects must have an adequate dataset available for calculating and reporting PK parameter | 129.5 (18)

20. Secondary Outcome: Accumulation Ratio (Rac) on Day 71
Description: Accumulation ratio was calculated from AUCinf at last dose/AUCinf at first dose, where AUCinf is defined as area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf). On Day 71, 3 participants in cohort 1 had reportable Rac values.
Time Frame: 0, 1, 4, hours post-dose on Day 71
Population: All participants randomized and treated who had at least 1 of the PK parameters of interest were analyzed. On Day 71, 3 participants in cohort 1 had reportable Rac values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1 PF-06342674 1 mg/kg | Cohort 2 PF-06342674 3 mg/kg | Cohort 4 PF-06342674 6 mg/kg | Cohort 3 PF-06342674 8 mg/kg
Number analyzed (Participants) | 8 | 8 | 2 | 8
Ratio | 1.115 (48) | 1.532 (28) | NA (NA) — Parameters not reported because less than 3 participants had reportable values, which failed to meet the Pfizer standard that at least 3 subjects must have an adequate dataset available for calculating and reporting PK parameter | 1.355 (19)

ADVERSE EVENTS:
Arm/Group | Placebo | PF-06342674 1 mg/kg | PF-06342674 3 mg/kg | PF-06342674 6 mg/kg | PF-06342674 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 1/9 | 0/5 | 0/8
Other Adverse Events (participants affected / at risk) | 5/7 | 6/8 | 6/9 | 4/5 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | PF-06342674 1 mg/kg (N=8) | PF-06342674 3 mg/kg (N=9) | PF-06342674 6 mg/kg (N=5) | PF-06342674 8 mg/kg (N=8)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | PF-06342674 1 mg/kg (N=8) | PF-06342674 3 mg/kg (N=9) | PF-06342674 6 mg/kg (N=5) | PF-06342674 8 mg/kg (N=8)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 1 | 1 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 1 | 1
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 1 | 0 | 0 | 1 | 1
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Epstein-Barr virus antibody positive (Investigations) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 2 | 0 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.